CLINICAL TRIAL: NCT05629351
Title: Prevalence of Sedentary Lifestyle, Pre-hypertension, and Obesity Among Healthy Young Adults
Brief Title: Prevalence of Sedentary Lifestyle, Pre-hypertension, and Obesity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Sumaya Shalabi, Principal investigator, Istanbul Saglik Bilimleri University
Other Study IDs: Saglikbilimleriuni
Record Dates: First submitted 2022-11-11; First posted 2022-11-29 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Health, Subjective; Healthy
Keywords: pre-hypertension; sedentary lifestyle; obesity; risk factors
MeSH Terms: conditions — Prehypertension; Sedentary Behavior; Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Group — Demographic Data (Blood pressure, subcutaneous fat tissue, height, waist and hip circumference, and body weight, BMI (body mass index) and double product)
  International Physical Activity Questionnaire (IPAQ)
  Godin-Shephard Leisure-Time Physical Activity Questionnaire
  The Dutch Eating Behavior Questionnaire
  Pittsburg Sleep Quality Questionnaire
  Perceived Stress Scale and Beck Depression Scale

SUMMARY:
Hypertension has been a serious problem among people from different ages in the last few decades, so by taking this in consideration we decided to search for specific risk factors that cause hypertension in young healthy adults, and to achieve that we are looking for pre-hypertension, obesity, and sedentary lifestyle among this group by using different scale tools and questionnaires.

DETAILED DESCRIPTION:
Hypertension has been a serious issue worldwide and there is a wide variety of content in literature regarding its risks, treatment modalities, and disease course. In this study, it was aimed to investigate the "pre-hypertension" state, which is the pre-step of hypertension, and to find its risk in young adults. While screening literature we found the incidence of pre-hypertension to be between 17% and 49% in individuals aged 18-30 years. However, study methods have generally been limited to blood pressure and anthropometric measurements. In our study, a holistic research will be carried out with different scales and questionnaires by enriching the method part.

The aim of this study is to determine the incidence of prehypertension, sedentary life and obesity in healthy young adults aged 18-25, and then to determine the relationship between these risk factors. 382 young adults will be included in this study. Blood pressure will be measured with a sphygmomanometer, subcutaneous fat tissue with a caliper, height with a height measurement device, waist and hip circumference with a tape measure, and body weight with a scale, BMI (body mass index) and double product will be recorded according to the data received by doing specific calculations. Participant's physical activity status will be evaluated with the International Physical Activity Scale and Leisure Activity Scale, dietary habits with the Dutch Eating Habits Questionnaire, sleep status with the Pittsburg Sleep Quality Questionnaire, and psychosocial status with the Perceived Stress Scale and Beck Depression Scale.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subjects

Exclusion Criteria:

* Smoker Subjects
* Alcohol drinker Subjects
* Subjects who use drugs that affect blood pressure

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Health young adult Subjects whose age between 18 to 25, female and male, and are willing to volunteer to this research
Sampling Method: Probability Sample
Enrollment: 382 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | baseline
  Systolic and Diastolic pressures are measured with a sphygmomanometer
Blood pressure | After 5 minutes from baseline
  Systolic and Diastolic pressures are measured with a sphygmomanometer
Blood pressure | After 10 minutes from baseline
  Systolic and Diastolic pressures are measured with a sphygmomanometer
Subcutaneous fat tissue | baseline
  Subcutaneous fat tissue is measured with a caliper in three regions (Biceps, Triceps, and abdomen)
Waist and Hip circumference | baseline
  waist and hip circumference is measured with a tape measure
Body weight | baseline
  body weight is measured with a scale

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | baseline
  he International Physical Activity Questionnaire (IPAQ) was developed to address these concerns by a group of experts in 1998 to facilitate surveillance of physical activity based on a global standard. The IPAQ has since become the most widely used physical activity questionnaire, with two versions available: the 31 item long form (IPAQ-LF) and the 9 item short form (IPAQ-SF). The short form records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting.
Dutch Eating Behavior Questionnaire (DEBQ) | baseline
  The Dutch Eating Behavior Questionnaire (DEBQ), developed by van Strien et al., simultaneously measures all three types of overeating proposed in these theories. It consists of 33 items covering the domains emotional eating (13 items), external eating (10 items), and restraint (10 items). All items are answered on a 5-point Likert scale ranging from 1('never') to 5 ('very often'). The Dutch original version of the DEBQ has been found to have good psychometric properties regarding reliability, factor structure and predictive validity.
  Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behavior.Cronbach alpha coefficients were above the recommended cut-off values of 0.80 for adequate consistency , whereas the test-retest reliability remains good.
Godin-Shephard Leisure-Time Physical Activity Questionnaire (GLTEQ) | baseline
  The GLTEQ measures the frequency of strenuous, moderate, and mild leisure-time physical activity performed for periods of 15 min or more over a usual week. Recently, a new scoring method has been proposed for generating an overall GLTEQ score that aligns with current recommendations for physical activity and the dose. The health contribution score (HCS) is based on only strenuous and moderate physical activity and is computed by multiplying the frequencies of strenuous and moderate activities by 9 and 5 metabolic equivalent of task (METs), respectively, and then adding the resultant scores. The HCS ranges between 0 and 98 and is converted into one of three categories, namely, insufficiently active (i.e., score <14 units that is the equivalent of <7 kcal/kg/week), moderately active (i.e., score between 14 and 23 units that is the equivalent of between 7 and 13.9 kcal/kg/week), and active (i.e., score ≥24 units that exceeds 13.9 kcal/kg/week).
The Perceived Stress Scale | baseline
  The Perceived Stress Scale (PSS-10) is a 10-item questionnaire originally developed by Cohen et al. (1983) widely used to assess stress levels in young people and adults aged 12 and above. It evaluates the degree to which an individual has perceived life as unpredictable, uncontrollable and overloading over the previous month.
  The questions ask about feelings and thoughts during the last month. In each case, respondents are asked how often they felt a certain way on a five-point scale from 'never' to 'very often'. Answers are then scored as follow: Never = 0 Almost never = 1 Sometimes = 2 Fairly often = 3 Very often = 4 To calculate a total PSS score, responses to the four positively stated items (items 4, 5, 7 and 8) first need to be reversed (i.e. 0 => 4; 1 => 3; 2 => 2; 3 => 1; 4 => 0).
  The PSS score is then obtained by summing across all items. Higher scores indicate higher levels of perceived stress.
Beck Depression Inventory II | baseline
  The Beck Depression Inventory II (BDI-II) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. The BDI has been developed in different forms, including several computerized forms, a card form the 13-item short form and the more recent BDI-II by Beck, Steer & Brown, 1996. The BDI takes approximately 10 minutes to complete, although clients require a fifth - sixth grade reading level to adequately understand the questions. There is a four-point scale for each item ranging from 0 to 3. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Cut-off score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Pittsburg Sleep Quality Questionnaire | baseline
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.
  Scores for each question range from 0 to 3. However PSQI minimum score is 0, maximum Score is 21 . TOTAL point < 5 associated with good sleep quality TOTAL > 5 associated with poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, ASST. Prof, Principal Investigator — Istanbul Saglik Bilimleri Universty; Seyedehatefeh Taghvatalab, Study Chair — Istanbul Saglik Bilimleri Universty; İlmiye Aktolgali, Study Chair — Istanbul Saglik Bilimleri Universty; Betul Kuzu, Study Chair — Istanbul Saglik Bilimleri Universty
Locations (1):
- Istanbul Saglik Bilimleri Universty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No